CLINICAL TRIAL: NCT03083626
Title: The Effects of Water Temperature on the Cold Pressor Test in Patients With Opioid-Induced Hyperalgesia in Comparison to Healthy Controls
Brief Title: The Effects of Water Temperature on the Cold Pressor Test
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-1378
Record Dates: First submitted 2017-03-07; First posted 2017-03-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Narcotic abuse; Opioid related disorders; Opiate substitution treatment; Buprenorphine; Pregabalin; Methadone
MeSH Terms: conditions — Chronic Pain; Narcotic-Related Disorders; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prescription opioid abusers: Patients 21-65 years old taking suboxone or methadone, currently experiencing chronic pain, not taking any opioid analgesic medication for painful condition on a regular basis, not have any current psychiatric or neurological illnesses, not have a history of heart disease in order to be healthy enough to complete the cold pressor test.
  Interventions: Other: Cold pressor test
- Healthy control participants: Patients 21-65 years old not taking suboxone or methadone, not experiencing chronic pain, not taking any opioid analgesic medication for painful condition on a regular basis, not have any current psychiatric or neurological illnesses, not have a history of heart disease in order to be healthy enough to complete the cold pressor test.
  Interventions: Other: Cold pressor test

INTERVENTIONS:
Other: Cold pressor test — The cold pressor test is a procedure used for examining pain threshold and tolerance by subjects placing their forearm in an ice bath. Each participant will take the CPT at 1 °C, 5°C, and 9°C. The first CPT will always be at 1 °C, to ensure participants tolerate the ice bath at the standard temperature. The order of the subsequent CPT at 5°C and 9°C, will be randomized to control for differential carry over effects. Participants will be instructed to say "Pain" when pain is initially detected (threshold). Then they will be asked to keep the immersed limb in the container until the pain can no longer be tolerated and say "Stop" and remove the arm from the water when tolerance is reached.

SUMMARY:
This current study is intended to be completed under the umbrella of the current GHUCCTS IRB- approved study "Opioid-Induced Hyperalgesia In Prescription Opioid Abusers: Effects of Pregabalin" (Lyrica study) (PRO00000669). In this proposed study, 10 healthy male, 10 healthy female participants and 5 male, 5 female OIH participants (from the parent Lyrica study), who are prescription opioid abusers with chronic pain currently taking Suboxone, will be asked to take the cold pressor test at 1, 5, and 9 degrees Celsius and to report the time at which pain has completely gone away following each test. The purpose of this study is to examine how the water temperature of the cold pressure test might affect the participants' response (i.e., the participants pain threshold and pain tolerance) and to see if there is a difference in how each participation group is affected.

DETAILED DESCRIPTION:
Since the 1940s, the cold pressor test (CPT) has been used experimentally as a pain induction method due to its reliability, cost effectiveness and minimal production of side effects. In the CPT, a patient is asked to place his or her hand and forearm in an ice bath until the pain is too great to remain in the water. Researchers have employed the CPT to test a wide range of pain management techniques, including medications, cognitive- based therapies, or acupuncture, as well as to explore pain perception. The CPT has been performed on a variety of participants, including adolescents, drug abusers, and those suffering from chronic back pain.

In their classic 1989 paper, Walsh and colleagues developed the normative model of the CPT demonstrating that variations in response are dependent upon age, sex and ethnicity. In 2004, however, Mitchell et al. discovered that the water temperature of the CPT also plays a crucial role in the pain tolerance time of the subjects, noting that a temperature variation of 4°C produced significantly different results for the same subject. While the Mitchell investigations improved upon the standard for the proper CPT technique, as seen implemented in the works of Rash and Campbell, their discoveries were based on healthy individuals.

Researchers have explored the CPT responses of patients with an altered pain perception, such as patients with Opioid-Induced Hyperalgesia (OIH), in comparison to healthy controls, demonstrating greater sensitivity in OIH patients. What has not been studied is the effect of temperature on CPT response in OIH patients. Further, the CPT has been shown to have a relatively lengthy recovery time averaging around 10 minutes; however, the recovery time for hypersensitive patients, such as OIH patients, has yet to be studied.

As an extension of the work of Mitchell and colleagues, the proposed research will assess the effects of temperature difference and recovery time of the CPT on patients with OIH in comparison to healthy normal control patients. This work is a sub-study of a larger study, Opioid-Induced Hyperalgesia In Prescription Opioid Abusers: Effects of Pregabalin (PRO00000669), conducted by principal investigator Dr. Peggy Compton. The goal of the parent study is to evaluate the ability of pregabalin to diminish chronic low back or arthritic pain and OIH in a sample of prescription opioid abusers (POAs) opioid therapy. This current study is not assigning specific interventions to study subjects. Healthy control and OIH participants will complete all study measures in a single two-hour study session.

ELIGIBILITY:
Inclusion Criteria:

* Between 21 and 65 years old
* On suboxone or methadone for at least ten days
* Currently experiencing chronic low back or arthritis pain

Exclusion Criteria:

* Be on any opioid analgesic
* Have a neurological or psychiatric illness (i.e., schizophrenia, Raynaud's disease, urticaria, stroke) that would affect pain responses
* Have an abnormal screening EKG, history of heart disease, stroke, liver or kidney disease or acute hepatitis, or currently have a pacemaker or uncontrolled high blood pressure.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 10 prescription opioid abusers with chronic low back or arthritis pain and stable on opioid therapy (on methadone or buprenorphine) will be enrolled in the study. Meeting the same inclusion exclusion criteria of the prescription opioid abusers (except treatment methadone or buprenorphine), a total of 20 male and female healthy controls will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Improved Pain Threshold Response | 1 two-hour study session
  In a well-described sample of prescription opioid abusers and healthy control subjects, the cold pressor test will be administered to examine how long it takes for a subject to start feeling pain when they immerse their forearm in the cold water (measured in seconds).
Improved Pain Tolerance Response | 1 two-hour study session
  In a well-described sample of prescription opioid abusers and healthy control subjects, the cold pressor test will be administered to examine how long subjects' can withstand feeling pain when they immerse their forearm in the cold water (measured in seconds).
Improved Pain Recovery Response | 1 two-hour study session
  In a well-described sample of prescription opioid abusers and healthy control subjects, the cold pressor test will be administered to examine how long it takes for subjects' to recover from the pain they experienced when they had their forearm immersed in the cold water (measured in seconds).

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahles, T. A., Blanchard, E. B., &Leventhal, H. (1983). Cognitive control of pain: Attention to the sensory aspects of the cold pressor stimulus. Cognitive Therapy and Research, 7(2), 159-177.
- [Background] Bellar D, Kamimori GH, Glickman EL. The effects of low-dose caffeine on perceived pain during a grip to exhaustion task. J Strength Cond Res. 2011 May;25(5):1225-8. doi: 10.1519/JSC.0b013e3181d9901f. PMID 21522070
- [Background] Brands AEF, Schmidt AJM. Learning processes in the persistence behavior of chronic low back pain patients with repeated acute pain stimulation. Pain. 1987 Sep;30(3):329-337. doi: 10.1016/0304-3959(87)90021-2. PMID 2959899
- [Background] Chang YP, Compton P. Management of chronic pain with chronic opioid therapy in patients with substance use disorders. Addict Sci Clin Pract. 2013 Dec 16;8(1):21. doi: 10.1186/1940-0640-8-21. PMID 24341916
- [Background] Chu LF, Clark DJ, Angst MS. Opioid tolerance and hyperalgesia in chronic pain patients after one month of oral morphine therapy: a preliminary prospective study. J Pain. 2006 Jan;7(1):43-8. doi: 10.1016/j.jpain.2005.08.001. PMID 16414554
- [Background] Compton MA. Cold-pressor pain tolerance in opiate and cocaine abusers: correlates of drug type and use status. J Pain Symptom Manage. 1994 Oct;9(7):462-73. doi: 10.1016/0885-3924(94)90203-8. PMID 7822886
- [Background] Compton P. Pain tolerance in opioid addicts on and off naltrexone pharmacotherapy: a pilot study. J Pain Symptom Manage. 1998 Jul;16(1):21-8. doi: 10.1016/s0885-3924(98)00035-9. PMID 9707654
- [Background] Edens, J. L., & Gil, K. M. (1995). Experimental induction of pain: Utility in the study of clinical pain. Behavior Therapy, 26(2), 197-216.
- [Background] Hellstrom B, Lundberg U. Pain perception to the cold pressor test during the menstrual cycle in relation to estrogen levels and a comparison with men. Integr Physiol Behav Sci. 2000 Apr-Jun;35(2):132-41. doi: 10.1007/BF02688772. PMID 11021338
- [Background] Lee M, Silverman SM, Hansen H, Patel VB, Manchikanti L. A comprehensive review of opioid-induced hyperalgesia. Pain Physician. 2011 Mar-Apr;14(2):145-61. PMID 21412369
- [Background] Mitchell LA, MacDonald RA, Brodie EE. Temperature and the cold pressor test. J Pain. 2004 May;5(4):233-7. doi: 10.1016/j.jpain.2004.03.004. PMID 15162346
- [Background] Pomerleau OF, Turk DC, Fertig JB. The effects of cigarette smoking on pain and anxiety. Addict Behav. 1984;9(3):265-71. doi: 10.1016/0306-4603(84)90018-2. PMID 6496202
- [Background] Radtke T, Eser P, Kriemler S, Saner H, Wilhelm M. Adolescent blood pressure hyperreactors have a higher reactive hyperemic index at the fingertip. Eur J Appl Physiol. 2013 Dec;113(12):2991-3000. doi: 10.1007/s00421-013-2735-3. PMID 24077645
- [Background] Walsh NE, Schoenfeld L, Ramamurthy S, Hoffman J. Normative model for cold pressor test. Am J Phys Med Rehabil. 1989 Feb;68(1):6-11. doi: 10.1097/00002060-198902000-00003. PMID 2917058
- [Background] Wolf S, Hardy JD. STUDIES ON PAIN. OBSERVATIONS ON PAIN DUE TO LOCAL COOLING AND ON FACTORS INVOLVED IN THE "COLD PRESSOR" EFFECT. J Clin Invest. 1941 Sep;20(5):521-33. doi: 10.1172/JCI101245. No abstract available. PMID 16694857